CLINICAL TRIAL: NCT01730261
Title: Online Emotional Regulation Group Treatment for Individuals With Traumatic Brain Injury (TBI)
Brief Title: Online Emotional Regulation Group Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1256-3; HSM 12-00760; IF1435434
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Traumatic Brain Injury; Executive Dysfunction; Emotional Dysregulation
Keywords: Traumatic Brain Injury; TBI; Executive Dysfunction; Emotional Regulation; Problem Solving; Self-regulation; Cognitive Rehabilitation; Metacognitive Strategies; Cognitive-behavioral therapy; Online Therapy; Group therapy; Group videoconference; Telehealth; Telerehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Emotional Regulation; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online Emotional Regulation Treatment (Experimental): Participants will receive 24 treatment sessions, with baseline, post-treatment screening and follow-up screening, and bi-weekly assessments
  Interventions: Behavioral: Online Emotional Regulation Treatment

INTERVENTIONS:
Behavioral: Online Emotional Regulation Treatment — Emotional Regulation Training (EmReg) is a cognitive-behavioral approach which aims to increase awareness, and self-monitoring of affective states to improve self-regulation. EmReg combines didactic and experiential training, and emphasizes skill acquisition and generalization through examination of incidents of emotional dysregulation in one's life and completion of homework assignments. The treatment is divided into two phases: knowledge provision and practice facilitation. During the knowledge provision phase participants are introduced to the objectives and the main concepts of the treatment, to increase their familiarity with the terminology, and to the emotional regulation skills they acquire during the practice facilitation phase. During the practice facilitation phase participants receive training in emotional regulation skills, which they practice in-session with the guidance of the therapist and feedback from the group, as well as out-of-session as homework assignments.
  Other Names: Emotional Regulation Training (EmReg)

SUMMARY:
This study will examine the feasibility of online delivery of emotional regulation training to individuals with TBI with emotional dysregulation. 80 subjects with significant emotional dysregulation will be enrolled and will receive 24 60-minute emotional regulation sessions twice a week for 12 weeks, delivered online in group modality. Attendance and compliance will be tracked, and outcomes will be monitored using online data collection methods. Treatment satisfaction and participant subjective experience will also be assessed.

DETAILED DESCRIPTION:
This study will examine the feasibility of online delivery of emotional regulation training to individuals with Traumatic Brain Injury who also have emotional dysregulation. 80 subjects with significant emotional dysregulation will be enrolled and will receive 24 60-minute emotional regulation sessions twice a week for 12 weeks, delivered online via a group meeting software. Study participation will last 28 weeks: 4 weeks of baseline, 12 weeks of treatment (24 sessions) and 12 weeks of follow-up. Assessments will be conducted at each of four timepoints: T1 (baseline), T2 (pre-treatment assessment), T3 (end-of-treatment assessment) and T4 (follow-up assessment). In addition, a subset of the measures will be administered bi-weekly for the duration of the study. Assessments will consist of a variety of measures designed to measure executive functioning, problem solving skills, and quality of life. All assessments will be completed online, using a web-based data collection. Attendance and treatment compliance will be tracked, and outcomes will be monitored using online data collection methods. Treatment satisfaction and participant subjective experience (including technical difficulties that make access to web-delivered treatment impossible) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Documented TBI of any severity and being at least 6 months post injury
* Presence of executive dysfunction, manifested as self-reported difficulties with emotional and behavioral self-regulation, operationalized as endorsement of 25% or more of the symptoms on the Difficulties in Emotion Regulation Scale (DERS, Gratz & Roemer, 2004).
* Currently aged 18 or older
* English speaking
* At least low average intellectual functioning, operationalized as a minimum Verbal IQ score of 80 on the Wechsler Abbreviated Scale of Intelligence
* Ownership of and relative facility with use of a computer, webcam, and microphone
* Access to a broadband internet connection at sufficiently high speed to allow videoconference

Exclusion Criteria:

* DSM-IV-TR diagnosis of alcohol or substance abuse within past 6 months
* DSM-IV-TR of psychosis within past 6 months
* High suicidality, operationalized as a score of 17 or higher on the Mini International Neuropsychiatric Interview (M.I.N.I., Sheehan et al., 2008)

Participation in this study will not preclude participation in other treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale(DERS) | up to 28 weeks
  36-item self-report questionnaire that focuses on emotional awareness, acceptance, ability to control impulsivity, and flexible use of strategies

SECONDARY OUTCOMES:
The Brain Injury Rehabilitation Trust Regulation of Emotions Questionnaire (BREQ) | up to 28 weeks
  32 item self-report questionnaire assessing deficits in emotion regulation, developed specifically to assess emotional dysregulation related to TBI
Problem Solving Inventory | up to 28 weeks
  35-item self-report questionnaire assessing problem solving capability
Social Problem Solving Inventory-Revised: Short Form | up to 28 weeks
  25-item self-report questionnaire assessing problem solving in everyday living
Positive Affect Negative Affect Scale | up to 28 weeks
  20-item self-report measure of positive and negative affect within a specified time frame
Satisfaction with Life Scale | T1 (baseline)
  5- item measure of global satisfaction with life
Satisfaction with Life Scale | T2 (week 4)
  5- item measure of global satisfaction with life
Satisfaction with Life Scale | T3 (week 16)
  5- item measure of global satisfaction with life
Satisfaction with Life Scale | T4 (week 28)
  5- item measure of global satisfaction with life
Satisfaction with Therapy and Therapist Scale | T3 (week 16)
  12-item scale that assesses satisfaction with treatment and therapist
Satisfaction with Therapy and Therapist Scale | T4 (week 28)
  12-item scale that assesses satisfaction with treatment and therapist
Treatment Compliance | up to 28 weeks
  therapist's ratings of participant on each of the following areas at each session: attendance, participation, homework completion, skill acquisition, skill generalization, ease of use of technology, and interpersonal behavior

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Brain Injury Research Center at Icahn School of Medicine at Mount Sinai, New York, New York, United States